CLINICAL TRIAL: NCT00748345
Title: Pharmacokinetics of Caspofungin in Burn Patients
Acronym: Caspo-brûlés
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070601
Record Dates: First submitted 2008-07-31; First posted 2008-09-08 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-07

CONDITIONS: Thermal Injury
Keywords: Caspofungin,; burn patients,; pharmacokinetics,; optimal dose,; antifungal treatment
MeSH Terms: interventions — Caspofungin; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Caspofungin (drug)
  Interventions: Drug: Caspofungin (drug)

INTERVENTIONS:
Drug: Caspofungin (drug) — pharmacokinetics of caspofungin in burn patients after a single usual dose (70 mg i.v.), in order to determine the optimal dose in this population
  Other Names: pharmacokinetics of caspofungin in burn patients

SUMMARY:
Drug pharmacokinetics of antimicrobial agents is significantly altered in the burn patients. Additionally, burn patient population exhibits a wide inter- and intrapatient variation in drug handling. Several investigations carried out in burn patients treated with e.g. fluconazole showed the requirement to increase daily dose in comparison with healthy volunteers. However, no pharmacokinetic data are available of caspofungin in the burn population. The aim of this investigation is to investigate pharmacokinetics of caspofungin in burn patients after a single usual dose (70 mg i.v.), in order to determine the optimal dose in this population.

DETAILED DESCRIPTION:
The aim of this investigation is to investigate pharmacokinetics of caspofungin in burn patients after a single usual dose (70 mg i.v.). Blood samples are drawn just before administration and 0.25, 0.5,1 1.5, 3, 6, 12, 24, 48, 72, 96 and 120 hours after administration. Caspofungin plasma concentrations are measured by liquid-chromatography spectrometry mass tandem.The primary end-points are :

* area under the curve of caspofungin plasma concentrations over 24 hours
* mean peak level and trough concentration (24 hours after dosing)

The secondary end-points are :

* mean total clearance
* mean distribution volume These parameters will be compared to those usually observed in non burn patients. The optimal dose in burn patients is the dose achieving an exposure similar to that in non burn patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 60 years old
* burn surface : 20-60% total body surface area
* delay of injury time : 8-15 days
* lack of fungal infection
* delay of hospitalization : > 5 days
* written informed consent
* last biological picture in 24 hours before inclusion

Exclusion Criteria:

* survival inferior to 5 days
* surgical intervention planned in the next five days following inclusion
* moderate or severe hepatic impairment according to Child Plug B > 9
* pregnancy
* allergy to caspofungin or excipients (saccharose, mannitol and frozen acetic acid)
* patient already included in other study
* concomitant administration of CYP450 inducers : rifampicin, efavirenz, phenobarbital, phenytoin, carbamazepine
* withdrawal of consent
* event (during the first 48 hours following administration) susceptible to modify pharmacokinetic parameters
* Investigator decision
* no social security insurance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
area under the curve of caspofungin plasma concentrations over 24 hours mean peak level and trough concentration (24 hours after dosing) | 18 months

SECONDARY OUTCOMES:
mean total clearance | 18 months
mean distribution volume | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Vinsonneau, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin, Paris, France